CLINICAL TRIAL: NCT01827826
Title: Translating the Diabetes Prevention Project (DPP) in a Health Maintenance Organization (HMO) Setting
Brief Title: Call-2-Health: Preventing Type II Diabetes
Acronym: C2H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 184802-16
Record Dates: First submitted 2012-09-11; First posted 2013-04-10 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Intervention; Telephone; Diabetes; Prevention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): Participants assigned to the intervention group worked with the study interventionist over the phone to reduce their risk for developing Diabetes Mellitus, Type 2. The intervention lasted for 24 weeks, with weekly phone calls for the first 12 weeks and 4 maintenance calls over the second 12 weeks. Study measurements were taken at baseline, 12 weeks, 24 weeks, and 52 weeks. After 24 weeks, the investigators randomly divided the intervention group in half. The first group did not receive any more phone calls from the interventionist. The second group continued to receive monthly 20-minute phone calls from the interventionist. At 52 weeks post-baseline participants from both groups had their labs drawn, wore a pedometer for 3 days, and called in with a self-reported weight.
  Interventions: Behavioral: Telephonic intervention to prevent Diabetes Mellitus, Type 2
- Control (No Intervention): Participants randomized into this group did not receive any intervention, although they were encouraged to follow-up with their doctor and follow through with usual clinical care.

INTERVENTIONS:
Behavioral: Telephonic intervention to prevent Diabetes Mellitus, Type 2 — Participants assigned to the intervention group received a total of 16 phone calls from the study interventionist over 24 weeks. The first 12 weeks was the intervention phase and calls were made weekly. The second 12 weeks was the maintenance phase and calls were made every 3 weeks. After 24 weeks, the investigators continued to follow this group for 52 weeks post-randomization, allowing half of the group to continue to receive monthly maintenance calls while the other half received no further calls. The study interventionist used behavior modification techniques to encourage intervention group participants to adopt healthy eating and exercise habits so that improvement might be seen in fasting glucose, glycated hemoglobin (HbA1c), weight, and waist/hip measurements.
  Arms: Intervention

SUMMARY:
It is estimated that 30 million U.S. adults will have type 2 diabetes by 2050. Contributing to this national trend is the obesity epidemic. Three randomized trials have demonstrated that intensive behavioral interventions can prevent or delay the onset of diabetes. The purpose of this pilot study is to inform a future randomized, controlled Phase III trial of a population-based, telephonic, exercise and weight loss intervention to translate the findings of the Diabetes Prevention Program into practice. The telephonic intervention will be compared to usual care (30 participants in each group). The investigators will deliver the intervention in 12 weekly, 20-minute calls, with four subsequent maintenance calls, for a total of 16 calls over 24 weeks. Study outcomes will be measured at baseline and at 12 and 24 weeks.

For this planning grant the investigators do not have an overall hypothesis. The investigators' goal is to develop and test whether it is possible to do exercise and weight loss

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 40-74
* Receives primary care at Group Health Central, Rainier, or Poulsbo clinics in the greater Seattle area
* Can walk for more than 10 minutes
* Fasting plasma glucose (FPG) 105-125 mg/dl or glycolated hemoglobin (HbA1C) 5.7-6.4
* Body Mass Index (BMI) 25 kg/m2 or greater

Exclusion Criteria:

* Type 1 or 2 diabetes
* FPG > 125 mg/dl or < 105mg/dl at screening blood draw
* HbA1C > 6.4 or < 5.7 at screening blood draw
* Systolic blood pressure > 210 mmHg at the baseline clinic visit
* Exercise ≥ 30 minutes/day, at least five days a week
* Current participation in another structured weight loss treatment program or another intervention study
* Severe concurrent disease
* Unavailable for the 24-week study period
* Unable to read or speak English
* Pregnant or planning to become pregnant.
* Mentally or legally incapacitated such that informed consent cannot be obtained.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-07; Primary Completion 2011-10 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Program feasibility: Uptake | Baseline
  Measured by the number of people who consent to be in the study compared to the number who were eligible
Program feasibility: Attendance | 12 weeks
  Measured by the number of participants who return for their 12 week clinic visit
Program feasibility: Attendance | 24 weeks
  Measured by the number of participants who return for their 24 week clinic visit
Program feasibility: Attendance | 52 weeks
  Measured by the number of participants who complete their 52 week assignments (3 day pedometer, self-reported weight, fasting blood draw)

SECONDARY OUTCOMES:
Fasting glucose | Baseline, 12 weeks, 24 weeks, 52 weeks
  Measured via a fasting blood draw
Waist circumference | Baseline, 12 weeks, 24 weeks
  in centimeters
Blood pressure | Baseline, 12 weeks, 24 weeks
  Measured using an automated clinical blood pressure monitor (Brand name: Omron, Model number HEM-907XL)
Healthy eating habits | Baseline, 12 weeks, 24 weeks
  Assessed using the Food Frequency Questionnaire
Weight loss | Baseline, 12 weeks, 24 weeks, 52 weeks
  Weight measured in kilograms
Changes in activity | Baseline, 12 weeks, 24 weeks, 52 weeks
  Measured using the Modifiable Activity Questionnaire (MAQ)
Glycated hemoglobin (A1C) | Baseline, 12 weeks, 24 weeks, 52 weeks
  Measured via a fasting blood draw
Total cholesterol (TC) | Baseline, 12 weeks, 24 weeks, 52 weeks
  Measured via a fasting blood draw
High density lipoprotein (HDL) | Baseline, 12 weeks, 24 weeks, 52 weeks
  Measured via a fasting blood draw
Low density lipoprotein (LDL) | Baseline, 12 weeks, 24 weeks, 52 weeks
  Measured via fasting blood draw.
Body Mass Index (BMI) | Baseline, 12 weeks, 24 weeks, 52 weeks
Physical activity level | Baseline, 12 weeks, 24 weeks, 52 weeks
  Participants wore a blinded pedometer for 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Newton, PhD, Principal Investigator — Group Health Research Institute
Locations (1):
- Group Health Research Institute, Seattle, Washington, United States